CLINICAL TRIAL: NCT01136330
Title: Cardiac and Respiratory Prognostic Factors in Patients With Myotonic Dystrophy Type 1
Brief Title: DM1 Heart Registry - DM1 Respiratory Registry
Acronym: DM1-Heart-R
Status: Completed | Type: Observational
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Principal Investigator, Karim WAHBI, Karim WAHBI MD,PHD., Institut de Myologie, France
Other Study IDs: AFM-13286
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Myotonic Dystrophy
Keywords: Myotonic dystrophy; Prognosis; Sudden death; Respiratory failure
MeSH Terms: conditions — Myotonic Dystrophy; Death, Sudden; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Myotonic dystrophy type 1 (DM1) is the most frequent neuromuscular disease in adults. DM1 patients have an impaired prognosis (mean age of death <60 years) due to cardiac and respiratory complications.

Our primary objective was to identify cardiac and respiratory prognostic factors in DM1.

DETAILED DESCRIPTION:
1. Patients with genetically proven DM1 who were admitted in Pitié Salpêtrière Hospital from 2000 and 2010 will be identified. These patients systematically underwent neurological, cardiac and respiratory investigations.
2. Baseline medical and genetic information will be entered in a dedicated database, including cardiac and respiratory investigations.
3. The occurence of severe cardiac and respiratory adverse events will also be collected.
4. Statistical analysis will be performed to look for correlations between baseline patient characteristics and cardiac or respiratory adverse events during follow up.

ELIGIBILITY:
Inclusion Criteria:

* DM1 mutation (>50 CTG repeats)
* Age > 18 years

Exclusion Criteria:

* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Myotonic dystrophy type 1
Sampling Method: Non-Probability Sample
Enrollment: 914 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Duboc, MD,PhD, Study Director — APHP
Locations (1):
- Pitié Salpêtrière Hospital, Paris, Île-de-France Region, France

REFERENCES:
- [Derived] Chong-Nguyen C, Wahbi K, Algalarrondo V, Becane HM, Radvanyi-Hoffman H, Arnaud P, Furling D, Lazarus A, Bassez G, Behin A, Fayssoil A, Laforet P, Stojkovic T, Eymard B, Duboc D. Association Between Mutation Size and Cardiac Involvement in Myotonic Dystrophy Type 1: An Analysis of the DM1-Heart Registry. Circ Cardiovasc Genet. 2017 Jun;10(3):e001526. doi: 10.1161/CIRCGENETICS.116.001526. PMID 28611030
- [Derived] Wahbi K, Babuty D, Probst V, Wissocque L, Labombarda F, Porcher R, Becane HM, Lazarus A, Behin A, Laforet P, Stojkovic T, Clementy N, Dussauge AP, Gourraud JB, Pereon Y, Lacour A, Chapon F, Milliez P, Klug D, Eymard B, Duboc D. Incidence and predictors of sudden death, major conduction defects and sustained ventricular tachyarrhythmias in 1388 patients with myotonic dystrophy type 1. Eur Heart J. 2017 Mar 7;38(10):751-758. doi: 10.1093/eurheartj/ehw569. PMID 27941019
- [Derived] Wahbi K, Algalarrondo V, Becane HM, Fressart V, Beldjord C, Azibi K, Lazarus A, Berber N, Radvanyi-Hoffman H, Stojkovic T, Behin A, Laforet P, Eymard B, Hatem S, Duboc D. Brugada syndrome and abnormal splicing of SCN5A in myotonic dystrophy type 1. Arch Cardiovasc Dis. 2013 Dec;106(12):635-43. doi: 10.1016/j.acvd.2013.08.003. Epub 2013 Oct 17. PMID 24140416
- [Derived] Wahbi K, Meune C, Porcher R, Becane HM, Lazarus A, Laforet P, Stojkovic T, Behin A, Radvanyi-Hoffmann H, Eymard B, Duboc D. Electrophysiological study with prophylactic pacing and survival in adults with myotonic dystrophy and conduction system disease. JAMA. 2012 Mar 28;307(12):1292-301. doi: 10.1001/jama.2012.346. PMID 22453570